CLINICAL TRIAL: NCT05598060
Title: Preoperative Stereotactic Body Radiotherapy (SBRT) Followed by Hepatectomy for Centrally Located Hepatocellular Carcinoma: a Prospective, Single-center, Phase I Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0743
Record Dates: First submitted 2022-10-18; First posted 2022-10-28 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-09

CONDITIONS: Centrally Located Hepatocellular Carcinoma; Stereotactic Body Radiotherapy; Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant stereotactic body radiation therapy followed by hepatectomy (Experimental): Experimental: Phase1(Cohort 1): neoadjuvant stereotactic body radiation therapy (24Gy/3Fr) followed by hepatectomy Experimental: Phase1(Cohort 2): neoadjuvant stereotactic body radiation therapy (30Gy/3Fr) followed by hepatectomy Experimental: Phase1(Cohort 3): neoadjuvant stereotactic body radiation therapy (36Gy/3Fr) followed by hepatectomy
  Interventions: Radiation: Neoadjuvant stereotactic body radiation therapy (Multiple ascending dose) followed by hepatectomy for centrally located hepatocellular carcinoma.

INTERVENTIONS:
Radiation: Neoadjuvant stereotactic body radiation therapy (Multiple ascending dose) followed by hepatectomy for centrally located hepatocellular carcinoma. — Neoadjuvant stereotactic body radiation therapy (Multiple ascending dose) followed by hepatectomy for centrally located hepatocellular carcinoma.

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth prevalent malignancy worldwide. Although surgical excision is considered the standard treatment for resectable HCC, a high rate of postoperative recurrence was observed after partial hepatectomy, with a marginal recurrence rate up to 30%. Narrow margin resection may be the most appropriate procedure for centrally located HCC because the premise for survival is the conservation of more normal liver parenchyma. Unfortunately, narrow margin resection has been reported to contribute to poor survival outcomes. However, no (neo)adjuvant therapy before (or after) hepatectomy is generally considered to be effective in reducing post-operative recurrence.

Radiotherapy (RT) has been well used in many solid malignant tumors as an (neo)adjuvant to surgical treatment, including HCC. SBRT has shown encouraging rates of local control for HCC. Compared with standard fractionation radiation, SBRT can achieve more precise delivery of high-dose radiation beams to the lesion, obtaining a much smaller target volume. Meanwhile, it could be finished in a short period which can bring more convenience to patients. Recently, several study and randomized controlled trials revealed the survival benefit of adjuvant RT (IMRT and SBRT) in patients with HCC. However, there are still lack of exploration for the efficacy of neoadjuvant SBRT. This study is to analyze the safety of preoperative SBRT followed by hepatectomy for centrally located hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Confirmed diagnosis of HCC. The diagnosis can be established radiographically by the criteria of the American Association for the Study of the Liver (AASLD), or by histologic diagnosis from the core biopsy;
3. Centrally located hepatocellular carcinoma and medically fit to undergo surgery as determined by the Multiple Disciplinary Team (MDT);
4. BCLC stage A
5. No imaging evidence of direct invasion of stomach, duodenum, small intestine, large intestine or diaphragm of the intrahepatic lesions to be treated with radiotherapy;
6. Child-Pugh class A and B7;
7. ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1;
8. Willing to provide tissue from an excisional biopsy of a tumor lesion;
9. For patients with active HBV: HBV DNA < 2000 IU/mL during screening, and have initiated anti-HBV treatment at least 7 days prior to SBRT and willingness to continue anti-HBV treatment during the study;
10. Adequate organ and marrow function as defined below:

1)Marrow: absolute neutrophil count ≥1.5×109/L; platelets ≥50×109/L; hemoglobin ≥90g/L; 2)Liver: total bilirubin ≤3× institutional upper limit of normal (ULN); AST(aspartate aminotransferase) or ALT(alanine aminotransferase) ≤ 5× institutional ULN; albumin ≥29g/L; 3)Kidney: creatinine ≤ 1.5× institutional ULN or estimated glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2 (according to the Cockcroft-Gault formula); 11. Women of childbearing potential must be willing to use a highly effective method of contraception for the course of the study through 30 days after radiotherapy. Female patient of childbearing potential should have a negative serum pregnancy test before 72h of her first treatment. Sexually active males must agree to use an adequate method of contraception starting with the treatment through 4 months after radiotherapy.

Exclusion Criteria:

1. Have received local or systemic treatments in the past, including but not limited to TACE, immunotherapy, targeted therapy, radiotherapy, radiofrequency therapy, etc.;
2. Severe bleeding tendency or coagulation dysfunction within the previous 6 months;
3. Extrahepatic metastasis;
4. Prior abdominal irradiation;
5. Any major surgery within 1 months prior to enrolment;
6. Known history of active Bacillus Tuberculosis (TB)
7. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
8. Active infection requiring systemic therapy;
9. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy;
10. Known psychiatric or substance abuse disorders ;
11. Pregnant or breastfeeding;
12. Known history of human immunodeficiency virus (HIV: HIV 1/2 antibodies);
13. Received a live vaccine within 30 days before radiotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of radiotherapy followed by hepatectomy : Incidence of Treatment-Emergent Adverse events (CTCAE v5.0) | 3 months after resection
  Safety and tolerability of radiotherapy followed by hepatectomy

SECONDARY OUTCOMES:
Local recurrence free survival | from date of enrollment to date of first documented local recurrence. Assessed up to 12 months
  Local recurrence free survival
Progression free survival | from date of enrollment to the date of first documented progression. Assessed up to 12 months
  Progression free survival
Overall survival | from date of enrollment to the date of death from any cause. Assessed up to 12 months
  Overall survival
Time to Progress | from date of enrollment to the date of progress. Assessed up to 12 months
  Time to Progress
Quality of life by EORTC QLQ-C30 | through study completion, an average of 1 year
  Quality of life by EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Qichun Wei, MD/PhD, Study Director — Zhejiang University; Weilin Wang, MD/PhD, Study Director — Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China